CLINICAL TRIAL: NCT05378256
Title: Chemotherapy Induced Peripheral Neuropathy (CIPN) in Lymphoma : Longitudinal Follow up and Prognostic Factors.
Brief Title: Chemotherapy Induced Peripheral Neuropathy (CIPN) and Lymphoma Longitudinal Follow-up and Prognostic Factors
Acronym: NeuroTox-L
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2021-09
Record Dates: First submitted 2022-01-12; First posted 2022-05-18 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma; Peripheral Neuropathy
Keywords: Chemotherapy induced peripheral neuropathy; Nerve conduction study; Vincristine; lymphoma
MeSH Terms: conditions — Lymphoma; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical scales of CIPN (Other): Patients with lymphoma will be evaluated before chemotherapy (T1), after 4 cycles (T2), at the end of the chemotherapy treatment (If more than 4 cycles) (T3) and 6 month after the end of chemotherapy (T4).
  Interventions: Other: Clinical scales of CIPN

INTERVENTIONS:
Other: Clinical scales of CIPN — Patients with lymphoma will be evaluated before chemotherapy (T1), after 4 cycles (T2), at the end of the chemotherapy treatment (If more than 4 cycles) (T3) and 6 month after the end of chemotherapy (T4).

SUMMARY:
Vincristine-induced peripheral neuropathy, which is commonly a sensorimotor neuropathy, remains a major complication of lymphoma patients treated with R-CHOP. The investigators propose a clinical, electrophysiological and biological follow up of patients treated by vincristine for lymphoma to determine the factors implied in VIPN occurrence.

DETAILED DESCRIPTION:
Patients with lymphoma will be evaluated before chemotherapy (T1), after 4 cycles (T2), at the end of the chemotherapy treatment (If more than 4 cycles) (T3) and 6 month after the end of chemotherapy (T4).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of indolent or aggressive B/T NHL confirmed by biopsy and requiring chemotherapy after PCR decision including vincristine, RCHOP/CHOP protocol or CHOEP
* Accept to participate in the study
* Age > 18 year
* Able and willing to provide informed consent
* Affiliated to a social security system

Exclusion Criteria:

* Life-threatening emergency requiring chemotherapy in extreme urgency
* Neuro-meningeal damage at diagnosis
* Protected person (under guardianship or curators)
* Person under court protection
* Pregnant or breastfeeding woman
* Persons deprived of liberty by judicial or administrative decision
* Persons under forced psychiatric care
* Persons admitted to a health or social institution for purposes other than research
* Persons unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Nerve conduction parameters | Before Chemotherapy first cure
  Nerve conduction study (NCS) with standard NCS of the tibial and peroneal motor, sural, sural dorsal, superficial peroneal, median, ulnar, and radial sensory nerves. ENMG study will be bilateral at lower limb and only left side at upper limb. T-Reflex and F-waves will be used to assess proximal nerve function.
Nerve conduction parameters | Immediately after 4th Chemotherapy course
  Nerve conduction study (NCS) with standard NCS of the tibial and peroneal motor, sural, sural dorsal, superficial peroneal, median, ulnar, and radial sensory nerves. ENMG study will be bilateral at lower limb and only left side at upper limb. T-Reflex and F-waves will be used to assess proximal nerve function.
Nerve conduction parameters | Immediately at the end of all the Chemotherapy courses
  Nerve conduction study (NCS) with standard NCS of the tibial and peroneal motor, sural, sural dorsal, superficial peroneal, median, ulnar, and radial sensory nerves. ENMG study will be bilateral at lower limb and only left side at upper limb. T-Reflex and F-waves will be used to assess proximal nerve function.
Nerve conduction parameters | 6 months after the end of all the cures
  Nerve conduction study (NCS) with standard NCS of the tibial and peroneal motor, sural, sural dorsal, superficial peroneal, median, ulnar, and radial sensory nerves. ENMG study will be bilateral at lower limb and only left side at upper limb. T-Reflex and F-waves will be used to assess proximal nerve function.

SECONDARY OUTCOMES:
Longitudinal study of the evolution of markers of neuropathy | Before Chemotherapy first cure
  The evolutionary follow-up will be done from NCI-CTC (National Cancer Institute-Common Toxicity Criteria) score (ranging from 0 - 4). Higher score mean a worse outcome.
Longitudinal study of the evolution of markers of neuropathy | Before Chemotherapy first cure
  The evolutionary follow-up will be done from the TNS (Total Neuropathy Score) scale which is based on symptoms, signs and basic instrumental evaluations and provides a much larger range of scoring values (0 - 40) than NCI-CTC scale, thus allowing the severity of CIPN to be graded more precisely. The TNS has so far been used to assess the neurotoxicity of various CIPN-relevant chemotherapeutic agents, and its results are clearly correlated with the clinically relevant results of NCI-CTC scale, which are commonly used by oncologists. Higher scores mean a worse outcome.
Longitudinal study of the evolution of markers of neuropathy | Before Chemotherapy first cure
  The evolutionary follow-up will be done from the DN4 scale which is a pain scale (ranging from 0 to 10) where 0 equals to no pain and 10 to maximum pain
Longitudinal study of the evolution of markers of neuropathy | Before Chemotherapy first cure
  The evolutionary follow-up will be done from the EORTC QOL-CIPN20 which is a quality of life scale (ranging from 0-80) where the lower score correspond to less symptoms and the highest score correspond to higher symptoms
Sudoscan (dysautonomic function) | Before Chemotherapy first cure
  Sudoscan performs a quantitative evaluation of sweat gland function based on an electrochemical reaction between sweat chlorides and electrodes in contact with the hands and feet using reverse iontophoresis and chronoamperometry
Gait parameters using FeetMe device | Before Chemotherapy (T1)
  The quantified evaluation of the subjects' walking will be carried out instrumentally over a 10-meter course using the FeetMe.
  FeetMeR Monitor insole (FeetMe, Paris, France) is a new wearable medical device (class Im) combining plantar pressure sensors, accelerometers, and gyroscopes.
Biological dosages | Before Chemotherapy (T1)
  Immunological factors (IL-6, IL-1b, TNF-a, IL-33, IL-10, CXCL1, CX3CL1)
Biological dosages | Before Chemotherapy (T1)
  Markers of peripheral nervous system damage (Claudine-5, Occludine, VEGF (Vascular Endothelial Growth Factor), BDNF (Brain-Derived Neurotrophic Factor)) will be mesured
Vincristin dosage | 1/4 hour after ending of each infusion
  Vincristin dosage will be performed at each infusion

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AUZOU, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR Orléans, Orléans, France

REFERENCES:
- [Background] Argyriou AA, Bruna J, Marmiroli P, Cavaletti G. Chemotherapy-induced peripheral neurotoxicity (CIPN): an update. Crit Rev Oncol Hematol. 2012 Apr;82(1):51-77. doi: 10.1016/j.critrevonc.2011.04.012. Epub 2011 Sep 10. PMID 21908200
- [Background] Caccia MR, Comotti B, Ubiali E, Lucchetti A. Vincristine polyneuropathy in man. A clinical and electrophysiological study. J Neurol. 1977 Aug 18;216(1):21-6. doi: 10.1007/BF00312811. PMID 72789
- [Background] Casey EB, Fullerton PM, Jelliffe AW. Vincristine neurotoxicity: a clinical and electrophysiological study of eighteen patients. Clin Sci. 1970 Apr;38(4):23P-24P. doi: 10.1042/cs038023pb. No abstract available. PMID 5428794
- [Background] Casey EB, Jellife AM, Le Quesne PM, Millett YL. Vincristine neuropathy. Clinical and electrophysiological observations. Brain. 1973;96(1):69-86. doi: 10.1093/brain/96.1.69. No abstract available. PMID 4348690